CLINICAL TRIAL: NCT04708327
Title: Randomized, Single-Blind Study to Evaluate the Pharmacokinetics, Biomarkers, Safety and Tolerability of STAT-205 in Adult Patients With Mild COVID 19 Who Are at High Risk of Disease Progression
Brief Title: Single-Blind Study of STAT-205 in Mild COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cytocom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST205-101-002
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Dosing Period 1: Placebo (five capsules) Dosing Period 2: Placebo (one capsule)
  Interventions: Drug: STAT-205
- STAT-205 (Experimental): Dosing Period 1: 22.5 mg STAT-205 (five 4.5 mg capsules) Dosing Period 2: 4.5 mg STAT-205 (one capsule)
  Interventions: Drug: STAT-205

INTERVENTIONS:
Drug: STAT-205 — naltrexone hydrochloride capsules 4.5 mg each

SUMMARY:
This is a randomized, single blind, study. Males and females meeting inclusion criteria who have symptoms of mild COVID-19 and in whom a positive PCR result for SARS-CoV-2 is obtained may be enrolled to the study treatment within 72 hours of the positive PCR result. Eligible patients are those considered to be at high risk for COVID-19 disease progression. This includes patients ≥ 65 years of age or with any one or more of certain medical conditions including: cancer, COPD, cardiovascular disease, immunocompromised state resulting from solid organ transplant, obesity, sickle cell disease, history of smoking, and diabetes.

DETAILED DESCRIPTION:
Eligible patients will be randomized, 1:2, to either placebo or STAT-205. Randomization will be stratified by site. STAT-205 treatment will include an initial 5-day dosing period (period 1) of 22.5 mg QD, to be followed by a second dosing period (period 2) of 4.5 mg QD to complete 30 days of dosing. Patients randomized to placebo will receive placebo QD. Blood samples for pharmacokinetic analysis and measurement of inflammatory biomarkers will be collected from patients on day 1, day 6, day 15 and day 30. Patients will be seen in the clinic on days 1, 6, 15, and 30. Patients will be contacted via telephone for follow up on day 60 and on. each post treatment day through Day 60. The telephone visit should occur at approximately the same time each day. During the telephone visits, the presence and severity of COVID-19 symptoms that were recorded at Baseline will be queried, and any new symptoms will be recorded. During the daily telephone visits, patients will also be queried for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 at the time of informed consent
2. Able to understand and provide informed consent in either English or Spanish
3. At high risk for COVID-19 disease progression by fulfilling at least ONE of the following criteria at Screening:

   1. Age ≥65 years
   2. Has a diagnosis of chronic pulmonary disease requiring daily treatment (e.g. COPD, chronic persistent asthma, cystic fibrosis, chronic bronchitis)
   3. Has a diagnosis of chronic heart disease
   4. Has a diagnosis of diabetes (type 1 or type 2) requiring oral therapy and/or insulin therapy
   5. Has hypertension requiring at least one oral medication for treatment
   6. Has a body mass index (BMI) of ≥33 kg/m2
   7. Has an immunocompromising disease (e.g. HIV infection with CD4 count < 200 cells/mm3)
   8. Is immunocompromised due to daily treatment with ≥20 mg of prednisone or equivalent
   9. Has received a solid organ transplant
   10. Has any chronic condition that, in the opinion of the investigator, places the patient at increased risk for progression of COVID-19
4. Documentation of positive diagnostic test for SARS-CoV-2 (confirmed by PCR assay or other approved diagnostic test) performed with a sample from nares or saliva, collected within 7 days of the Screening visit.
5. Is symptomatic for COVID-19 for no more than 7 days prior to the Screening visit
6. Has a WHO Clinical Progression Scale (WHOb 2020) score of either '2' or '3' at Screening and Randomization
7. Has at least one of the following symptoms at the Screening visit that are new in onset, or if present by history, has worsened during the 7 days prior to Screening:

   · fever, chills, myalgia, arthralgia, headache, fatigue, cough, sore throat, nasal congestion, nausea, vomiting, diarrhea, anosmia or dysosmia, ageusia or dysgeusia
8. If female of child-bearing potential, must agree to use of 2 forms of contraception from Screening to end of the study. Males must agree to use 2 forms of contraception from screening to the end of the study if their partners are of childbearing potential. Acceptable methods of birth control which must be used together are:

   1. Oral or injectable contraceptive and condom, or
   2. IUD and condom, or
   3. Diaphragm with spermicide and condom.
9. Agrees to participate in all in-person visits and remote or home visits as required by the protocol and to provide updated contact information, as necessary.

Exclusion Criteria:

1. Has a WHO Clinical Progression Scale (WHOb 2020) score of '4' or higher at Screening or Enrollment
2. Previous hypersensitivity or allergic reactions to naltrexone
3. Women who are pregnant or lactating or expecting to become pregnant
4. Drugs of abuse screen positive for opiates
5. Patients with history of moderate to severe renal impairment (estimated creatinine clearance < 50 mL/min) or hepatic impairment (Child-Pugh C)
6. Serum ALT or AST value > 3 times the ULN at Screening
7. Serum creatinine value > 2 times the ULN at Screening, or requires renal dialysis
8. Hematology results at Screening showing any one of the following: WBC <2000 cells/mm3 or platelet count <100,000 cells/mm3 or hemoglobin <8.5 Gm/dL
9. Currently receiving chronic daily opioid therapy
10. Use of tocilizumab or other immunomodulator therapy directed to treatment or prevention of COVID-19
11. History of active substance abuse within the 2 years prior to Screening
12. Participation in another clinical trial investigating a treatment for COVID-19
13. Currently hospitalized or under immediate consideration for hospitalization (for any medical reason) at the Screening visit
14. At Screening, has new onset of dyspnea (shortness of breath) or, if previously diagnosed with a chronic lung condition, the severity of dyspnea has increased over patient's historical baseline condition (increased dyspnea should be present continually and not intermittent)
15. Measurement of oxygen saturation at Screening is < 94% on ambient room air
16. Shares a household with a patient currently enrolled in this protocol
17. Patients who refuse biomarker blood draws

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-05 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who demonstrate progression of COVID-19 disease | Day 1 to Day 30
  Progression of COVID-19 disease based on the WHO clinical progression scale (WHOb2020)

CONTACTS AND LOCATIONS:
Overall Officials: George Azar, MD, Principal Investigator — Clinical Research Center of Florida; Jennifer Veltman, MD, Principal Investigator — Loma Linda University
Locations (2):
- United States (2):
  - Loma Linda University, Loma Linda, California
  - Clinical Research Center of Florida, Pompano Beach, Florida

IPD SHARING:
Plan to Share IPD: No